CLINICAL TRIAL: NCT02203734
Title: Massage to Reduce Intrauterine Artery Resistance, Prematurity and Low Birthweight
Brief Title: Massage To Improve Uterine Artery Blood Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Miguel Diego (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Miguel Diego, Research Associate Professor, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20080617; R21HD069872-01A1 (NIH)
Record Dates: First submitted 2013-11-28; First posted 2014-07-30 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Pregnancy; Depression
Keywords: Pregnancy; Depression; Massage
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Moderate Pressure Massage (Experimental): Moderate Pressure Massage Therapy
  Interventions: Procedure: Moderate Pressure Massage
- Light Pressure Massage (Sham Comparator): Light Pressure Massage Therapy
  Interventions: Procedure: Light Pressure Massage

INTERVENTIONS:
Procedure: Moderate Pressure Massage — The massage therapy will begin with the mother in a side-lying position, with pillows positioned behind her back and between her legs for support. The massage is given in the following sequence and repeated twice (10 minutes on each side for 20 minutes total) on the following areas: 1) Head and neck: 2) Back: 3) Arms: and 4) Legs. The effective moderate pressure (measured by a pressure meter) is 8 db or a slight indentation in the skin.
  Arms: Moderate Pressure Massage
Procedure: Light Pressure Massage — The light pressure massage group will receive light pressure massage in contrast to the treatment group who will receive moderate pressure massage. As with moderate pressure massage, each session will begin with the mother in a side-lying position, with pillows positioned behind her back and between her legs for support. The massage is given in the following sequence and repeated twice (10 minutes on each side for 20 minutes total) on the following areas: 1) Head and neck: 2) Back: 3) Arms: and 4) Legs.
  Arms: Light Pressure Massage

SUMMARY:
This project will investigate the effects of massage therapy on depressed pregnant women. The investigators expect that massage therapy will improve blood flow from the mother to the fetus and reduce prematurity and depression.

DETAILED DESCRIPTION:
Prenatal depression has been associated with adverse neonatal outcomes including preterm birth and low birthweight. Potential underlying mechanisms for prenatal depression effects on prematurity and low birthweight involve the elevated sympathetic nervous system SNS and Hypothalamic Pituitary Adrenal HPA Axis function noted in depressed pregnant women. These may lead to increased uterine artery resistance and the resulting limited blood flow, oxygen and nutrients to the fetus. Moderate pressure massage therapy may reduce this problem in depressed pregnant women by decreasing SNS and HPA axis function, resulting in decreased uterine artery resistance, increased oxygen and nutrients to the fetus and lower prematurity and low birthweight. An alternative model being explored here is that moderate pressure massage may increase progesterone/estriol ratios, which counteract the negative cortisol effects on gestational age. Eighty pregnant women with depression symptoms will be recruited at approximately 20 weeks gestation and randomly assigned to a moderate pressure massage therapy or to a SHAM light pressure massage touch/attention control group. The women will receive 20-minute weekly massage therapy sessions from 20 to 30 weeks gestation. At 20 and 30 weeks gestation, depressed symptoms will be assessed using the CES-D, and saliva samples will be collected to assay alpha amylase as an SNS marker, cortisol as an HPA axis marker and progesterone and estriol levels. Maternal Doppler ultrasound will be conducted to assess the uterine artery resistance index as an estimate of uterine artery blood flow. Upon delivery, the mothers' medical charts will be reviewed to record gestational age and birthweight. The investigators are hypothesizing that the moderate pressure massage group will elicit an increase in progesterone/estriol ratios and decreases in alpha amylase and cortisol levels, which in turn will lead to reduced uterine artery resistance and a lower incidence of prematurity and low birthweight.

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated singleton pregnancy
* Depression
* < 20 weeks GA at recruitment

Exclusion Criteria:

* Pregnancy complications
* HIV
* Smoking, drug use

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change Doppler Ultrasound | First Day of Study and 10 Weeks After
  Change in Doppler Ultrasound to assess Uterine Artery Resistance Index values

SECONDARY OUTCOMES:
Change in CES-D | First Day of Study and 10 Weeks After
  Change in Depression Questionaire Scores
Change Saliva Samples | First Day of Study and 10 Weeks After
  Saliva samples to assess changes in cortisol and alpha amylase
Birth Outcome Data | Birth
  Obtain birth outcome data (Birthweight and Gestational age) from medical records after birth of baby

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami, Miami, Florida, United States

REFERENCES:
- See also: Touch Research Institute — http://www6.miami.edu/touch-research/